CLINICAL TRIAL: NCT07239921
Title: Disease Characteristics of Rapidly Progressive Coronary Artery Disease (R-CAD): A Case-control Study
Brief Title: Disease Characteristics of R-CAD
Status: Not yet recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, LiuZhenyu, Professor, Peking Union Medical College Hospital
Other Study IDs: K9096
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Coronary Artery Disease; Coronary Artery Disease Progression; Coronary Stenosis; Coronary Restenosis; Coronary Stent Occlusion; Myocardial Revascularization; Percutaneous Coronary Intervention
Keywords: Coronary Artery Disease; Coronary Stenosis; Coronary Restenosis; Myocardial Revascularization; Percutaneous Coronary Intervention; Disease Progression; Disease Attributes
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis; Coronary Restenosis; Disease Progression; Disease Attributes | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood samples will be retained for exploratory tests, including RNA sequencing, proteomics, and metabolomics, et al.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case Group: R-CAD patients
  Interventions: Diagnostic Test: Protocol-defined Examinations and Evaluations
- Control Group: NR-CAD patients
  Interventions: Diagnostic Test: Protocol-defined Examinations and Evaluations

INTERVENTIONS:
Diagnostic Test: Protocol-defined Examinations and Evaluations — Lab tests (blood and urine and stool routine tests, hepatic and renal and thyroid function tests, tests for metabolic markers, tests for cardiac biomarkers, thrombosis-related tests, rheumatology tests, tests for inflammation markers), electrocardiography, echocardiography, 6-minute walk test, vascular ultrasound, coronary angiography, optical coherence tomography (OCT), fibroblast activation protein inhibitor positron emission tomography/computed tomography (FAPI-PET/CT), photon-counting detector coronary computed tomography angiography (PCD-CCTA), tests for exploratory biomarkers.

SUMMARY:
The present case-control study is designed to investigate the disease characteristics of rapidly progressive coronary artery disease (R-CAD) by comparing the demographics, clinical features, lab results, imaging findings, and prior treatment between patients in the case group (approximately 34 patients with R-CAD) and those in the control group (approximately 18 patients with non-rapidly progressive coronary artery disease [NR-CAD]).

DETAILED DESCRIPTION:
The majority of coronary artery disease (CAD) is atherosclerotic coronary artery disease (AS-CAD), the pathological basis of which is atherosclerosis. Secondary prevention, including healthy life style and medical treatment, effectively controls the progression of AS-CAD. Coronary revascularization, including percutaneous coronary intervention (PCI) and coronary artery bypass graft (CABG) are the dominant treatment modalities to restore the patency and/or blood flow of the diseased coronary arteries.

A special type of CAD is identified in the investigators' clinical practice, which progresses rapidly and recurs frequently after PCI or CABG, and responds poorly to intensified secondary prevention for AS-CAD. The investigators name this special type of CAD with rapidly progressive coronary artery disease (R-CAD), which has significantly different clinical features from those of typical AS-CAD. The CAD without the above characteristics is named with non-rapidly progressive coronary artery disease (NR-CAD).

Currently, the disease characteristics of R-CAD remain unknown. It has been identified that a proportion of R-CAD patients demonstrate certain manifestations of inflammation, including positive inflammatory markers, or positive autoantibodies, or established diagnosis of chronic inflammatory diseases, or use of immunosuppressive therapy, whose R-CAD is named as inflammation-associated rapidly progressive coronary artery disease (IR-CAD). However, the rest of R-CAD patients demonstrate no manifestations of inflammation. Therefore, the present case-control study is designed to investigate the disease characteristics of the overall R-CAD patients by comparing the demographics, clinical features, lab results, imaging findings, and prior treatment between the case group (approximately 34 patients with R-CAD) and the control group (approximately 18 patients with NR-CAD).

Patients will be enrolled in the case group (R-CAD patients) of the present case-control study if they 1) have prior history of coronary revascularization (PCI or CABG); 2) received standard treatment for secondary prevention of AS-CAD after the latest coronary revascularization; 3) have evidence of rapidly progressive myocardial ischemia leading to hospitalization and/or coronary revascularization; 4) have angiographic evidence of rapidly progressive coronary lesions leading to myocardial ischemia.

Patients will be enrolled in the control group (NR-CAD patients) of the present case-control study if they 1) are 35 to 75 years old; 2) received standard treatment for secondary prevention of AS-CAD after the latest PCI which was performed 12±6 months ago; 3) do not have evidence of rapidly progressive myocardial ischemia leading to hospitalization and/or coronary revascularization; 4) do not have angiographic evidence of rapidly progressive coronary lesions leading to myocardial ischemia.

Once enrolled, patients in both groups will receive examinations and evaluations according to a clinical management protocol specifically designed for the clinical management of R-CAD patients. The information regarding the baseline characteristics and the results of examinations and evaluations, including demographics, clinical features, lab results, imaging findings, and prior treatment, will be collected and compared between the case group and the control group.

The primary endpoint is the rate of elevated erythrocyte sedimentation rate (ESR) or high-sensitivity C-reactive protein (hs-CRP).

ELIGIBILITY:
Inclusion Criteria:

Case Group (R-CAD patients):

1. 18 years of age or older, male or female.
2. Negative results of urine or blood pregnancy test for females with childbearing potential (not post-menopausal or surgically sterile).
3. Prior history of coronary revascularization (PCI or CABG).
4. Receiving standard treatment for secondary prevention of AS-CAD after the latest coronary revascularization.
5. Rapidly progressive myocardial ischemia leading to hospitalization and/or coronary revascularization:

   1. Typical symptoms of angina (Canadian Cardiovascular Society [CCS] classification III-IV) and non-invasive evidence of myocardial ischemia; and
   2. Occurred within 6 months of the latest ischemia-driven hospitalization and/or coronary revascularization.
6. Rapidly progressive coronary lesions leading to myocardial ischemia:

   1. Angiographic evidence of new-onset or worsened coronary de novo or restenotic lesions relevant to myocardial ischemia, and
   2. Occurred within 6 months of the latest ischemia-driven coronary angiography and/or revascularization.

Control Group (NR-CAD patients):

1. 35 to 75 years old*, male or female. (* Based on the age distribution characteristics of patients who have been diagnosed as R-CAD.)
2. Negative results of urine or blood pregnancy test for females with childbearing potential (not post-menopausal or surgically sterile).
3. Currently, at 12±6 months after the latest PCI.
4. Receiving standard treatment for secondary prevention of AS-CAD after the latest PCI.
5. Coronary angiography and/or optical coherence tomography (OCT) performed during the index hospitalization.
6. No evidence of rapidly progressive myocardial ischemia and coronary lesions, i.e., not fulfilling items 5) and 6) of the inclusion criteria for R-CAD.

Exclusion Criteria:

1. Receiving immunosuppressive therapy within 6 months.
2. Coronary restenosis due to mechanical factors (stent under-expansion, stent mal-apposition, stent rupture, et al).
3. Other moderate to severe heart diseases (congenital heart disease, valvular heart disease, myocarditis, cardiomyopathy, pericardial diseases, pulmonary hypertension, heart failure, arrhythmia, et al).
4. Active malignancy (diagnosed within 12 months or with ongoing requirement for treatment).
5. Vital organ failure.
6. Life expectancy < 1 year.
7. In pregnancy or breast-feeding, or with intention to be pregnant during the study period.
8. Risk of non-compliance (history of drug addiction or alcohol abuse, et al).
9. Previous enrollment in this study.
10. Participation in another study within 30 days.
11. Involvement in the planning and conduct of this study (applying to investigators, contract research organization staffs, study site staffs, et al).
12. Any condition, which in the opinion of the investigators, would make it unsuitable for the patient to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who fulfill the inclusion/exclusion criteria for R-CAD defined by the protocol of the present case-control study will be enrolled in the case group of the present case-control study.
  Patients who fulfill the inclusion/exclusion criteria for NR-CAD defined by the protocol of the present case-control study will be enrolled in the control group of the present case-control study.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Elevated ESR or hs-CRP | From 30 days before enrollment up to 14 days after enrollment, but before the initiation of immunosuppressive therapy.
  Percentage of patients with elevated ESR (> 15 mm/h for male or > 20 mm/h for female) or hs-CRP (≥ 2 mg/L).

SECONDARY OUTCOMES:
Positive autoantibodies | From 30 days before enrollment up to 14 days after enrollment, but before the initiation of immunosuppressive therapy.
  Percentage of patients with positive autoantibodies (anti-nuclear antibody [ANA], anti-neutrophil cytoplasmic antibody [ANCA], anti-endothelial cell antibody [AECA], lupus anticoagulant [LA], antiphospholipid antibody (APL) (anti-cardiolipin antibody [ACL], anti-beta2-glycoprotein 1 antibody [abeta2GP1]), anti-phosphatidylserine antibody [APSA], rheumatoid factor [RF], anti-cyclic citrullinated peptide antibody [anti-CCP], et al.).
Established diagnosis of chronic inflammatory diseases | Up to 14 days after enrollment
  Percentage of patients with established diagnosis of chronic inflammatory diseases (chronic infectious disease, autoimmune disease, other chronic inflammatory diseases, et al.).
Elevated ESR or hs-CRP, or positive autoantibodies | From 30 days before enrollment up to 14 days after enrollment, but before the initiation of immunosuppressive therapy.
  Percentage of patients with elevated ESR or hs-CRP, or positive autoantibodies.
Elevated ESR or hs-CRP, or positive autoantibodies, or established diagnosis of chronic inflammatory diseases | For elevated ESR or hs-CRP and positive autoantibodies: from 30 days before enrollment up to 14 days after enrollment, but before the initiation of immunosuppressive therapy; for established diagnosis of chronic inflammatory diseases: up to 14 days after
  Percentage of patients with elevated ESR or hs-CRP, or positive autoantibodies, or established diagnosis of chronic inflammatory diseases.

OTHER OUTCOMES:
Maximum standardized uptake value (SUVmax) | From 30 days before enrollment up to 14 days after enrollment, but before the initiation of immunosuppressive therapy.
  SUVmax based on fibroblast activation protein inhibitor positron emission tomography/computed tomography (FAPI-PET/CT).
Maximum target background ratio (TBRmax) | From 30 days before enrollment up to 14 days after enrollment, but before the initiation of immunosuppressive therapy.
  TBRmax based on fibroblast activation protein inhibitor positron emission tomography/computed tomography (FAPI-PET/CT).
Fat attenuation index (FAI) | From 30 days before enrollment up to 14 days after enrollment, but before the initiation of immunosuppressive therapy.
  FAI based on photon-counting detector coronary computed tomography angiography (PCD-CCTA).

CONTACTS AND LOCATIONS:
Overall Officials: Zhenyu Liu, M.D., Principal Investigator — Peking Union Medical College Hospital

IPD SHARING:
Plan to Share IPD: No